CLINICAL TRIAL: NCT00033657
Title: Randomized Phase II Study of Preoperative Combined Modality Paclitaxel / Cisplatin / RT or Irinotecan / Cisplatin / RT Followed by Postoperative Chemotherapy With the Same Agents in Operable Adenocarcinoma of the Esophagus
Brief Title: Radiation Therapy and Chemotherapy Before and After Surgery in Treating Patients With Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069309; U10CA021115 (NIH); E1201 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Platinum; Irinotecan; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisplatin / Irinotecan / Radiation therapy (Arm A) (Experimental): Days 1 - 35 : Concurrent radiation therapy (RT) and Cisplatin / Irinotecan Chemotherapy. Radiotherapy 45 Gy administered at 1.8 Gy per day, 5 days a week for 5 weeks. Cisplatin 30 mg/m² days 1, 8, 22, 29. Irinotecan 65 mg/m² days 1, 8, 22, 29. Chemotherapy should begin within 24 hours of start of radiotherapy
  Days 63 - 77 : Surgical Resection At least 28 days after surgical resection, begin adjuvant chemotherapy: cisplatin 30 mg/m² and irinotecan 65 mg/m² days 1 and 8 of three 3-week cycles
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Procedure: conventional surgery; Radiation: radiation therapy
- Paclitaxel / Cisplatin / Radiation therapy (Arm B) (Experimental): Days 1 - 35 : Concurrent radiation therapy (RT) and Paclitaxel/Cisplatin Chemotherapy. Radiotherapy 45 Gy administered at 1.8 Gy per day, 5 days a week for 5 weeks. Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29. Cisplatin 30 mg/m² days 1, 8, 15, 22, 29. Chemotherapy should begin within 24 hours of start of radiotherapy.
  Days 63 - 77 : Surgical Resection At least 28 days after surgical resection, begin adjuvant chemotherapy: paclitaxel 175 mg/m² and cisplatin 75 mg/m² day 1 of three 3-week cycles.
  Interventions: Drug: cisplatin; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — Days 1 - 35 : Cisplatin 30 mg/m² days 1, 8, 15, 22, 29
  Days 63 - 77 : cisplatin 30 mg/m² and irinotecan 65 mg/m² days 1 and 8 of three 3-week cycles
  Other Names: cis-platinum; platinum; Platinol; Platinol-AQ; DDP; CDDP; DACP; NSC 119875
Drug: irinotecan hydrochloride — Days 1 - 35 : Irinotecan 65 mg/m² days 1, 8, 22, 29
  Days 63 - 77 : irinotecan 65 mg/m² days 1 and 8 of three 3-week cycles
  Other Names: Camptothecin-11; CPT-11; Camptosar
  Arms: Cisplatin / Irinotecan / Radiation therapy (Arm A)
Drug: paclitaxel — Days 1 - 35 : Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29
  Days 63 - 77 : paclitaxel 175 mg/m² and cisplatin 75 mg/m² day 1 of three 3-week cycles
  Other Names: Taxol; NSC 125973
  Arms: Paclitaxel / Cisplatin / Radiation therapy (Arm B)
Procedure: conventional surgery — The type of resection (lvor-Lewis, Transhiatal, etc.) was left to the discretion of the operating surgeon. One lymph node dissection was required.
Radiation: radiation therapy — The total dose to the prescription point was 4500 cGy given in 25 fractions. The patient was treated with one fraction per day with all fields treated per day. 180 cGy was delivered to the isocenter. If the dose to the supraclavicular fossa (SCF) was less than 4500 cGy, a localized photon or electron boost was allowed in order to increase the SCF dose to 4500 cGy, specified at 3 cm depth from the anterior skin surface.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy before and after surgery may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of combining radiation therapy with two different chemotherapy regimens before and after surgery in treating patients who have esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the pathologic complete response rate in patients with adenocarcinoma of the esophagus or gastroesophageal junction treated with radiotherapy with pre- and post-operative cisplatin plus paclitaxel versus cisplatin plus irinotecan.
* Compare the survival outcome in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the tolerability of these adjuvant chemotherapy regimens after neoadjuvant chemoradiotherapy in these patients.
* Compare time to progression or recurrence in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG performance status (0 vs. 1) and stage of disease (T2-3, N0, M0 vs. T1-3, N0-1, M0 or M1A). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive neoadjuvant radiotherapy once daily, 5 days a week, for 5 weeks beginning on day 1 concurrently with neoadjuvant chemotherapy comprising cisplatin IV (Intravenous) over 2-3 hours followed by irinotecan IV over 30-60 minutes once daily on days 1, 8, 22, and 29. Four to six weeks after completion of neoadjuvant chemoradiotherapy, patients undergo surgical resection. A minimum of 4 weeks after resection, patients receive adjuvant chemotherapy comprising cisplatin and irinotecan as above on days 1 and 8. Treatment with adjuvant chemotherapy repeats every 3 weeks for 3 courses.
* Arm B: Patients receive neoadjuvant radiotherapy as in arm A concurrently with neoadjuvant chemotherapy comprising paclitaxel IV (Intravenous) over 1 hour followed by cisplatin IV over 2-3 hours once daily on days 1, 8, 15, 22, and 29. Patients then undergo surgical resection as in arm A. A minimum of 4 weeks after resection, patients receive adjuvant chemotherapy comprising paclitaxel IV over 3 hours followed by cisplatin as above on day 1. Treatment with adjuvant chemotherapy repeats every 3 weeks for 3 courses.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month, every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ACCRUAL: A total of 97 patients (50 on Arm A and 47 on Arm B) were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adenocarcinoma of the esophagus (20 cm below incisors) or gastroesophageal junction

  * Stage T2-3, N0, M0 OR
  * Stage T1-3, N0-1, M0 or M1A (celiac nodal metastasis)
* Tumor must be considered surgically resectable (T1-3, but not T4)
* Age>=18 years
* ECOG Performance status 0-1
* Adequate hematopoietic, hepatic, renal functions defined by the following within 4 weeks prior to randomization:
* Granulocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Prior curatively treated malignancy allowed if currently disease-free and survival prognosis is more than 5 years
* Fertile patients must use effective contraception
* Endoscopy with biopsy and dilation allowed

Exclusion Criteria:

* Tumor extends more than 2 cm into the cardia
* Pregnant or nursing
* Other concurrent illness that would preclude study therapy or surgical resection
* Concurrent filgrastim (G-CSF) during study radiotherapy
* Prior chemotherapy
* Prior radiotherapy
* Prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-08-15 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Kleinberg, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (23):
- United States (23):
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Kleinberg L, Powell ME, Forastiere AA, et al.: Survival outcome of E1201: An Eastern Cooperative Oncology Group (ECOG) randomized phase II trial of neoadjuvant preoperative paclitaxel/cisplatin/radiotherapy (RT) or irinotecan/cisplatin/RT in endoscopy with ultrasound (EUS) staged esophageal adenocarcinoma. [Abstract] J Clin Oncol 26 (Suppl15): A-4532, 2008.
- [Result] Kleinberg LR, Eapen S, Hamilton S, et al.: E1201: an Eastern Cooperative Oncology Group (ECOG) randomized phase II trial to measure response rate and toxicity of preoperative combined modality paclitaxel/cisplatin/RT or irinotecan/cisplatin/RT in adenocarcinoma of the esophagus. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-143, S80, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E1201 opened to accrual on May 21, 2002 and accrued its first patient on August 15, 2002. A total of 97 patients were accrued from 19 different participating sites.
Groups:
- Cisplatin / Irinotecan / RT (Arm A): Days 1 - 35 : Concurrent radiation therapy and Cisplatin / Irinotecan Chemotherapy. Radiotherapy 45 Gy administered at 1.8 Gy per day, 5 days a week for 5 weeks. Cisplatin 30 mg/m² days 1, 8, 22, 29. Irinotecan 65 mg/m² days 1, 8, 22, 29. Chemotherapy should begin within 24 hours of start of radiotherapy
  Days 63 - 77 : Surgical Resection At least 28 days after surgical resection, begin adjuvant chemotherapy: cisplatin 30 mg/m² and irinotecan 65 mg/m² days 1 and 8 of three 3-week cycles
- Paclitaxel / Cisplatin / RT (Arm B): Days 1 - 35 : Concurrent RT and Paclitaxel/Cisplatin Chemotherapy. Radiotherapy 45 Gy administered at 1.8 Gy per day, 5 days a week for 5 weeks. Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29. Cisplatin 30 mg/m² days 1, 8, 15, 22, 29. Chemotherapy should begin within 24 hours of start of radiotherapy.
  Days 63 - 77 : Surgical Resection At least 28 days after surgical resection, begin adjuvant chemotherapy: paclitaxel 175 mg/m² and cisplatin 75 mg/m² day 1 of three 3-week cycles.
Period: Neoadjuvant Chemotherapy
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B)
Started | 50 | 47
Eligible | 42 | 43
Eligible and Treated | 39 | 42
Completed | 36 | 36
Not Completed | 14 | 11
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — other complicating disease | 0 | 1
Not completed — Ineligible | 8 | 4
Not completed — Not started protocol therapy | 3 | 1
Period: Surgical Resection
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B)
Started | 36 | 36
Completed | 36 | 33
Not Completed | 0 | 3
Not completed — not complete resection | 0 | 3
Period: Adjuvant Chemotherapy
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B)
Started | 36 | 33
Completed | 18 | 16
Not Completed | 18 | 17
Not completed — Lack of Efficacy | 3 | 1
Not completed — Adverse Event | 7 | 10
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — alternative therapy | 1 | 0
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B) | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.7) | 59.9 (10.7) | 58.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 35 | 35 | 70
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: A patient would have achieved a pathologic complete response if no histopathological evidence of residual tumor is found in the resected esophageal specimen and nodal tissue.
Time Frame: approximately 1 month after completing all treatments, then every 3 months up to 2 years, every 6 months from 2-5 years of study entry and annually 6-10 years from study entry
Population: Eligible, treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B)
Number analyzed (Participants) | 39 | 42
percentage of participants | 15.4 [6.9 to 28.1] | 16.7 [8.1 to 29.0]

2. Secondary Outcome: Overall Survival Time
Description: Survival was measured from the date of randomization onto study to death from any cause.Patients who were still alive at the end of the study were censored at the last date of known alive. Median survival time was calculated in the 81 eligible and treated patients.
Time Frame: as for outcome 1
Population: Eligible, treated patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B)
Number analyzed (Participants) | 39 | 42
Months | 35.0 [19.5 to 67.7] | 21.0 [17.4 to 49.3]
Statistical Analysis 1: Comparison: Cisplatin / Irinotecan / RT (Arm A) vs Paclitaxel / Cisplatin / RT (Arm B); Test type: Superiority or Other; p = 0.48, Log Rank

3. Secondary Outcome: Recurrence-free Survival Time
Description: Recurrence-free survival is measured from the date of complete response to recurrence of the cancer. Patients without recurrence were censored at the last date of known recurrence-free. Median recurrence-free survival time was calculated in the eligible and treated patients.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cisplatin / Irinotecan / RT (Arm A) | Paclitaxel / Cisplatin / RT (Arm B)
Number analyzed (Participants) | 39 | 42
Months | 39.8 [13.3 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 12.4 [11.0 to 31.4]

ADVERSE EVENTS:
Time Frame: Reported 4-6 weeks after the end of pre-op chemotherapy/RT, (just prior to resection) and 4 weeks after the end of adjuvant chemotherapy
Groups:
- Neoadjuvant_Cisplatin / Irinotecan / RT (Arm A): Days 1 - 35 : Concurrent radiation therapy and Cisplatin / Irinotecan Chemotherapy. Radiotherapy 45 Gy administered at 1.8 Gy per day, 5 days a week for 5 weeks. Cisplatin 30 mg/m² days 1, 8, 22, 29. Irinotecan 65 mg/m² days 1, 8, 22, 29. Chemotherapy should begin within 24 hours of start of radiotherapy
  Days 63 - 77 : Surgical Resection At least 28 days after surgical resection, begin adjuvant chemotherapy: cisplatin 30 mg/m² and irinotecan 65 mg/m² days 1 and 8 of three 3-week cycles
- Neoadjuvant_Paclitaxel / Cisplatin / RT (Arm B): Days 1 - 35 : Concurrent RT and Paclitaxel/Cisplatin Chemotherapy. Radiotherapy 45 Gy administered at 1.8 Gy per day, 5 days a week for 5 weeks. Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29. Cisplatin 30 mg/m² days 1, 8, 15, 22, 29. Chemotherapy should begin within 24 hours of start of radiotherapy.
  Days 63 - 77 : Surgical Resection At least 28 days after surgical resection, begin adjuvant chemotherapy: paclitaxel 175 mg/m² and cisplatin 75 mg/m² day 1 of three 3-week cycles.
- Adjuvant_Cisplatin / Irinotecan / RT ( Arm A): Adjuvant chemotherapy toxicities in treated patients
Arm/Group | Neoadjuvant_Cisplatin / Irinotecan / RT (Arm A) | Neoadjuvant_Paclitaxel / Cisplatin / RT (Arm B) | Adjuvant_Cisplatin / Irinotecan / RT ( Arm A) | Adjuvant_Paclitaxel / Irinotecan / RT ( Arm B)
Serious Adverse Events (participants affected / at risk) | 32/47 | 30/46 | 20/31 | 15/27
Other Adverse Events (participants affected / at risk) | 47/47 | 46/46 | 30/31 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant_Cisplatin / Irinotecan / RT (Arm A) (N=47) | Neoadjuvant_Paclitaxel / Cisplatin / RT (Arm B) (N=46) | Adjuvant_Cisplatin / Irinotecan / RT ( Arm A) (N=31) | Adjuvant_Paclitaxel / Irinotecan / RT ( Arm B) (N=27)
Leukopenia (Investigations) | 17 | 16 | 15 | 6
Lymphopenia (Investigations) | 0 | 1 | 0 | 1
Neutropenia (Investigations) | 15 | 13 | 16 | 8
Thrombocytopenia (Investigations) | 1 | 1 | 1 | 0
Transfusion:PRBCS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0
Thrombosis/Embolism (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 5 | 2 | 2
Fever (General disorders) | 0 | 1 | 1 | 0
Weight loss (Investigations) | 1 | 1 | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 9 | 2 | 5 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 4 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dysphagia-esophageal radiation (Injury, poisoning and procedural complications) | 6 | 8 | 0 | 1
Mucositis due to radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 6 | 1 | 3
Vomiting (Gastrointestinal disorders) | 4 | 4 | 3 | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 1 | 5 | 3
Bilirubin increased (Investigations) | 1 | 0 | 1 | 0
AST increased (Hepatobiliary disorders) | 0 | 1 | 0 | 0
ALT increased (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 2
Infection w/o neutropenia (Infections and infestations) | 1 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dizziness/lightheadedness (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy-motor (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0 | 0
Neuropathic pain (Nervous system disorders) | 0 | 1 | 0 | 0
Pain due to radiation (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Pain-other (General disorders) | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0
Urinary electrolyte wasting (Renal and urinary disorders) | 0 | 1 | 0 | 0
Erectile impotence (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Dysphagia-pharyngeal radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant_Cisplatin / Irinotecan / RT (Arm A) (N=47) | Neoadjuvant_Paclitaxel / Cisplatin / RT (Arm B) (N=46) | Adjuvant_Cisplatin / Irinotecan / RT ( Arm A) (N=31) | Adjuvant_Paclitaxel / Irinotecan / RT ( Arm B) (N=27)
Anemia (Blood and lymphatic system disorders) | 38 | 40 | 28 | 22
Leukopenia (Investigations) | 44 | 41 | 27 | 17
Neutropenia (Investigations) | 35 | 24 | 23 | 9
Thrombocytopenia (Investigations) | 31 | 29 | 21 | 8
Edema (General disorders) | 1 | 4 | 1 | 0
Fatigue (General disorders) | 32 | 33 | 23 | 19
Weight loss (Investigations) | 19 | 17 | 15 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 13 | 10 | 14
Radiation dermatitis (Injury, poisoning and procedural complications) | 8 | 6 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 21 | 18 | 11 | 14
Constipation (Gastrointestinal disorders) | 10 | 12 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 12 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 7 | 4 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 4 | 1 | 2
Dysphagia-esophageal radiation (Injury, poisoning and procedural complications) | 18 | 21 | 3 | 2
Dysphagia-pharyngeal radiation (Injury, poisoning and procedural complications) | 7 | 2 | 1 | 0
Mouth dryness (Gastrointestinal disorders) | 3 | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 26 | 30 | 19 | 14
Stomatitis (Gastrointestinal disorders) | 3 | 8 | 0 | 0
Taste disturbance (Gastrointestinal disorders) | 9 | 15 | 8 | 10
Vomiting (Gastrointestinal disorders) | 20 | 16 | 10 | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 17 | 16 | 14 | 13
Alkaline phosphatase increased (Investigations) | 10 | 7 | 10 | 7
Bilirubin increased (Investigations) | 4 | 6 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 4 | 1 | 1
AST increased (Hepatobiliary disorders) | 5 | 9 | 2 | 3
ALT increased (Hepatobiliary disorders) | 17 | 17 | 5 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 9 | 3 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 6 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 4 | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 7 | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 9 | 2 | 1
Dizziness/lightheadedness (Nervous system disorders) | 5 | 11 | 2 | 2
Insomnia (Psychiatric disorders) | 4 | 2 | 1 | 2
Anxiety/agitation (Psychiatric disorders) | 3 | 4 | 1 | 3
Neuropathy-sensory (Nervous system disorders) | 4 | 7 | 3 | 12
Abonominal pain (Gastrointestinal disorders) | 8 | 7 | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2 | 1
Creatinine increased (Investigations) | 8 | 12 | 3 | 8
Dysuria (Renal and urinary disorders) | 1 | 3 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Inner ear/hearing imparied (Ear and labyrinth disorders) | 2 | 2 | 2 | 1
Hypotension (Vascular disorders) | 1 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No